CLINICAL TRIAL: NCT00177372
Title: Mifepristone and Misoprostol for the Treatment of Early Pregnancy Failure: a Pilot Clinical Trial
Brief Title: Mifepristone and Misoprostol for Fetal Demise
Acronym: MIMID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pittirb0409119
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Anembryonic Pregnancy; Gestation Abnormality; Intrauterine Fetal Demise Term
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Mifepristone 200 mg followed 24 hours later by misoprostol 800 mcg vaginally
  Interventions: Drug: mifepristone/misoprostol

INTERVENTIONS:
Drug: mifepristone/misoprostol — mifepristone 200 mg followed 24 hours later by misoprostol 800 mcg vaginally
  Other Names: Mifeprix/Cytotec

SUMMARY:
This is a pilot clinical trial to evaluate whether the medical management of early pregnancy failure with mifepristone and misoprostol is an effective and acceptable treatment. Subjects with early pregnancy failure receive mifepristone followed 24 hours later by vaginal misoprostol for medical management. Subjects then return on study day 3 for a repeat ultrasound to assess passage of pregnancy tissue. subjects who still have a gestational sac present at Day 3 receive a second dose of vaginal misoprostol. All subjects have a follow-up at Day 15, by phone for those who passed the pregnancy with the first dose of misoprostol, and in person for those who received a second dose. Questionnaires are administered at the beginning and end of the study to determine acceptability.

ELIGIBILITY:
Inclusion Criteria: healthy hemodynamically stable females with a non-viable pregnancy

-

Exclusion Criteria:

* orthostatic hypotension, contraindication to either mifepristone or misoprostol, treatment during current pregnancy to provide surgical or medical evacuation of the uterus, evidence of ovarian hyperstimulation syndrome, known or suspected pelvic infection,known or suspected clotting defect or receiving anticoagulants, cardiovascular disease, current breastfeeding, pregnancy with and IUD in situ, current participation in another clinical trial, prior participation in this trial, suspected or confirmed endometrial AV malformation, clinical indication requiring the karyotyping of products of conception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
to determine if medical management with mifepristone and misoprostol for early pregnancy failure is an effective and acceptable treatment | 1-2 weeks

SECONDARY OUTCOMES:
to evaluate if the treatment of early pregnancy failure with mifepristone and misoprostol is as effective as induced abortion with these medications | 1-2 weeks
to assess if mifepristone/misoprostol treatment is acceptable to patients with early pregnancy failure | 1-2 weeks
to assess the predictors/indicators for successful mifpristone/misoprostol treatment in patients with early pregnancy failure | 1-2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell D Creinin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schreiber CA, Creinin MD, Reeves MF, Harwood BJ. Mifepristone and misoprostol for the treatment of early pregnancy failure: a pilot clinical trial. Contraception. 2006 Dec;74(6):458-62. doi: 10.1016/j.contraception.2006.07.007. Epub 2006 Sep 7. PMID 17157102